CLINICAL TRIAL: NCT00908115
Title: Evaluation of Safety and Efficacy Through Post Market Surveillance for Infanrix™, the DTaP Mixed Vaccine
Brief Title: Post Market Surveillance for Infanrix™
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 208355/128
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Diphtheria; Acellular Pertussis; Tetanus
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Pentetic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Infanrix Group: Subjects received one dose of Infanrix™ at 2, 4 and 6 months of age (primary vaccination), one dose at 15-18 months of age (booster vaccination) and one dose at 4-6 years of age (booster vaccination).
  Interventions: Biological: GSK Biologicals' Infanrix™

INTERVENTIONS:
Biological: GSK Biologicals' Infanrix™ — Primary and booster vaccination according to vaccination schedule. Intramuscular injection
  Other Names: DTPa

SUMMARY:
The purpose of this study was to investigate the following questions through post-marketing surveillance:

* Unknown/Unexpected adverse events and the serious adverse events.
* The circumstances in which the adverse events occurred under the practical application.
* Factors considered to have influence on safety.
* Factors considered to have influence on efficacy.
* Miscellaneous - Facts about mechanism, efficacy and safety which were not clearly known due to the inherent problems of the drugs.

ELIGIBILITY:
Inclusion Criteria:

All children receiving Infanrix™ were eligible for this survey.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All children receiving Infanrix™ were eligible for this survey.
Sampling Method: Non-Probability Sample
Enrollment: 1258 (Actual)
Dates: Start 2003-08-01 (Actual); Primary Completion 2008-06-23 (Actual); Study Completion 2008-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=364

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 208355/128 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208355/128 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208355/128 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208355/128 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208355/128 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208355/128 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infanrix Group
Started | 1258
Completed | 1244
Not Completed | 14
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Arm/Group | Infanrix Group
Number analyzed (Participants) | 1258
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.0 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 615
  Male | 643

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: A serious adverse event is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Since the beginning of the study and during the entire study period (up to 6 years)
Measure: Number; unit: Subjects
Arm/Group | Infanrix Group
Number analyzed (Participants) | 1258
Subjects | 3

2. Primary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include induration, itching, pain, redness, and swelling. Solicited general symptoms assessed include anorexia, convulsions, cough, diarrhea, drowsiness, eruption, fever, irritability, and vomiting.
Time Frame: During the 4-week follow-up period after each dose
Population: Analysis was performed on the subjects who received the considered dose.
Measure: Number; unit: Subjects
Arm/Group | Infanrix Group
Number analyzed (Participants) | 877
Subjects
  Induration after Dose 1 (n=798) | 51
  Induration after Dose 2 (n=843) | 72
  Induration after Dose 3 (n=877) | 86
  Induration after Booster at 15-18 Months (n=88) | 19
  Induration after Booster at 4-6 Years (n=22) | 5
  Itching after Dose 1 (n=798) | 5
  Itching after Dose 2 (n=843) | 8
  Itching after Dose 3 (n=877) | 2
  Itching after Booster at 15-18 Months (n=88) | 8
  Itching after Booster at 4-6 Years (n=22) | 4
  Pain after Dose 1 (n=798) | 29
  Pain after Dose 2 (n=843) | 31
  Pain after Dose 3 (n=877) | 43
  Pain after Booster at 15-18 Months (n=88) | 13
  Pain after Booster at 4-6 Years (n=22) | 6
  Redness after Dose 1 (n=798) | 51
  Redness after Dose 2 (n=843) | 76
  Redness after Dose 3 (n=877) | 79
  Redness after Booster at 15-18 Months (n=88) | 22
  Redness after Booster at 4-6 Years (n=22) | 4
  Swelling after Dose 1 (n=798) | 26
  Swelling after Dose 2 (n=843) | 43
  Swelling after Dose 3 (n=877) | 51
  Swelling after Booster at 15-18 Months (n=88) | 20
  Swelling after Booster at 4-6 Years (n=22) | 5
  Anorexia after Dose 1 (n=798) | 41
  Anorexia after Dose 2 (n=843) | 40
  Anorexia after Dose 3 (n=877) | 31
  Anorexia after Booster at 15-18 Months (n=88) | 5
  Anorexia after Booster at 4-6 Years (n=22) | 0
  Convulsions after Dose 1 (n=798) | 1
  Convulsions after Dose 2 (n=843) | 1
  Convulsions after Dose 3 (n=877) | 2
  Convulsions after Booster at 15-18 Months (n=88) | 0
  Convulsions after Booster at 4-6 Years (n=22) | 0
  Cough after Dose 1 (n=798) | 21
  Cough after Dose 2 (n=843) | 18
  Cough after Dose 3 (n=877) | 20
  Cough after Booster at 15-18 Months (n=88) | 3
  Cough after Booster at 4-6 Years (n=22) | 0
  Diarrhea after Dose 1 (n=798) | 15
  Diarrhea after Dose 2 (n=843) | 15
  Diarrhea after Dose 3 (n=877) | 20
  Diarrhea after Booster at 15-18 Months (n=88) | 4
  Diarrhea after Booster at 4-6 Years (n=22) | 0
  Drowsiness after Dose 1 (n=798) | 47
  Drowsiness after Dose 2 (n=843) | 41
  Drowsiness after Dose 3 (n=877) | 38
  Drowsiness after Booster at 15-18 Months (n=88) | 5
  Drowsiness after Booster at 4-6 Years (n=22) | 1
  Eruption after Dose 1 (n=798) | 6
  Eruption after Dose 2 (n=843) | 7
  Eruption after Dose 3 (n=877) | 13
  Eruption after Booster at 15-18 Months (n=88) | 2
  Eruption after Booster at 4-6 Years (n=22) | 0
  Fever after Dose 1 (n=798) | 40
  Fever after Dose 2 (n=843) | 36
  Fever after Dose 3 (n=877) | 17
  Fever after Booster at 15-18 Months (n=88) | 6
  Fever after Booster at 4-6 Years (n=22) | 2
  Irritability after Dose 1 (n=798) | 90
  Irritability after Dose 2 (n=843) | 82
  Irritability after Dose 3 (n=877) | 74
  Irritability after Booster at 15-18 Months (n=88) | 9
  Irritability after Booster at 4-6 Years (n=22) | 1
  Vomiting after Dose 1 (n=798) | 20
  Vomiting after Dose 2 (n=843) | 13
  Vomiting after Dose 3 (n=877) | 13
  Vomiting after Booster at 15-18 Months (n=88) | 1
  Vomiting after Booster at 4-6 Years (n=22) | 0

3. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: An adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within the 31-day (Day 0-30) following vaccination.
Measure: Number; unit: Subjects
Arm/Group | Infanrix Group
Number analyzed (Participants) | 1258
Subjects | 144

ADVERSE EVENTS:
Time Frame: SAES were collected during the entire study period (Day 0 up to 6 years), Unsolicited AEs: within Day 0-30 and Solicited AEs during 4 weeks post vaccination periods. No unsolicited AEs with a frequency >5% were reported. Therefore the total number of participants at risk in Other AE section is the highest number of participants at risk analysed for solicited AEs (i.e. after Dose 3). PRI = primary; D1 = Dose 1; D2 = Dose 2; D3= Dose 3; BST = Booster ;15-18 Months = 15-18M; 4-6 Years = 4-6Y.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Infanrix Group
All-Cause Mortality (participants affected / at risk) | 0/1258
Serious Adverse Events (participants affected / at risk) | 3/1258
Other Adverse Events (participants affected / at risk) | 90/877
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix Group (N=1258)
Croup infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infanrix Group (N=877)
Induration PRI D1 (General disorders) | 51/798 — The number of subjects at risk is the total number of subjects that received the respective dose.
Induration PRI D2 (General disorders) | 72/843 — The number of subjects at risk is the total number of subjects that received the respective dose.
Induration PRI D3 (General disorders) | 86 — The number of subjects at risk is the total number of subjects that received the respective dose.
Redness PRI D1 (General disorders) | 51/798 — The number of subjects at risk is the total number of subjects that received the respective dose.
Redness PRI D2 (General disorders) | 76/843 — The number of subjects at risk is the total number of subjects that received the respective dose.
Redness PRI D3 (General disorders) | 79 — The number of subjects at risk is the total number of subjects that received the respective dose.
Swelling PRI D2 (General disorders) | 43/843 — The number of subjects at risk is the total number of subjects that received the respective dose.
Drowsiness PRI D1 (General disorders) | 47/798 — The number of subjects at risk is the total number of subjects that received the respective dose.
Irritability PRI D1 (General disorders) | 90/798 — The number of subjects at risk is the total number of subjects that received the respective dose.
Irritability PRI D2 (General disorders) | 82/843 — The number of subjects at risk is the total number of subjects that received the respective dose.
Irritability PRI D3 (General disorders) | 74 — The number of subjects at risk is the total number of subjects that received the respective dose.
Swelling PRI D3 (General disorders) | 51
Induration BST 15-18M (General disorders) | 19/88
Itching BST 15-18M (General disorders) | 8/88
Pain BST 15-18M (General disorders) | 13/88
Redness BST 15-18M (General disorders) | 22/88
Swelling BST 15-18M (General disorders) | 20/88
Induration BST 4-6Y (General disorders) | 5/22
Itching BST 4-6Y (General disorders) | 4/22
Pain BST 4-6Y (General disorders) | 6/22
Redness BST 4-6Y (General disorders) | 4/22
Swelling BST 4-6Y (General disorders) | 5/22
Anorexia PRI D1 (General disorders) | 41/798
Fever PRI D1 (General disorders) | 40/798
Anorexia BST 15-18M (General disorders) | 5/88
Drowsiness BST 15-18M (General disorders) | 5/88
Fever BST 15-18M (General disorders) | 6/88
Irritability BST 15-18M (General disorders) | 9/88
Fever BST 4-6Y (General disorders) | 2/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.